CLINICAL TRIAL: NCT07249684
Title: Effect of Myofascial Release and Static Stretching Along With Nighttime Bracing in Long-Term Relapse Prevention of Ponseti Treated Clubfoot
Brief Title: Myofascial Release And Static Stretching Along With Nighttime Bracing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Maryam Rehman MS-PT/02178
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Clubfoot Deformity
Keywords: Myofascial release; Static stretching; Clubfoot deformity; Ponseti Technique
MeSH Terms: conditions — Clubfoot | interventions — Myofascial Release Therapy; Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release (Experimental): The intervention protocol for the experimental group (group A) includes Direct myofascial release on calf muscle (gastrocnemius and soleus) and tibialis posterior muscle for 2 mints.
  Total 4 sessions per week for 4 weeks with a total of 16 sessions. Conventional therapy: conventional therapy includes gentle mobilization of subtalar and talocrural joint grade2 (5 reps in 1 set) and night time brace.
  Total 4 sessions per week for 4 weeks with a total of 16 sessions.
  Interventions: Other: Myofascial release
- static stretching (Experimental): intervention protocol for 2nd Experimental Group (Group B) includes static stretching of calf muscle (gastrocnemius and soleus and tibialis posterior (5 reps with 10 sec hold).
  Total 4 sessions per week for 4 weeks with a total of 16 sessions. conventional therapy: conventional therapy conventional therapy includes gentle mobilization of subtalar and talocrural joint grade 2 (5 reps in 1 set) and night time brace.
  Total 4 sessions per week for 4 weeks with a total of 16 sessions.
  Interventions: Other: Static Stretching

INTERVENTIONS:
Other: Myofascial release — The intervention protocol for the experimental group (group A) includes Direct myofascial release on calf muscle (gastrocnemius and soleus) and tibialis posterior muscle for 2 mints.
  Total 4 sessions per week for 4 weeks with a total of 16 sessions.
  Conventional therapy: conventional therapy includes gentle mobilization of subtalar and talocrural joint grade2 (5 reps in 1 set) and night time brace.
  Total 4 sessions per week for 4 weeks with a total of 16 sessions.
  Arms: Myofascial release
Other: Static Stretching — intervention protocol for 2nd Experimental Group (Group B) includes static stretching of calf muscle (gastrocnemius and soleus and tibialis posterior (5 reps with 10 sec hold).
  Total 4 sessions per week for 4 weeks with a total of 16 sessions. conventional therapy: conventional therapy conventional therapy includes gentle mobilization of subtalar and talocrural joint grade 2 (5 reps in 1 set) and night time brace.
  Total 4 sessions per week for 4 weeks with a total of 16 sessions.
  Arms: static stretching

SUMMARY:
The goal of this randomized controlled trial is to learn if Myofascial Release and Static Stretching combined with Nighttime Bracing can prevent long-term relapse of Ponseti-treated idiopathic clubfoot in children with idiopathic clubfoot. The main questions it aims to answer are:

Does the addition of Myofascial Release and Static Stretching to Nighttime Bracing reduce the rate of long-term relapse in Ponseti-treated clubfoot? Does this combined intervention improve long-term mobility and quality of life in children with idiopathic clubfoot?

Researcher will compare the group receiving Myofascial Release with night time bracing o the group receiving Static Stretching along with Nighttime to see the effect of both intervention reduces relapse rates and improves functional outcomes.

Participants will:

Receive Myofascial Release and Static Stretching therapy sessions Use Nighttime Bracing as prescribed Undergo follow-up assessments to evaluate relapse occurrence, mobility, and quality of life

DETAILED DESCRIPTION:
Clubfoot, or congenital talipes equinovarus, is a common congenital deformity occurring in 1 to 2 per 1,000 live births globally, with higher prevalence in males and certain populations. Defined by midfoot cavus, forefoot adducts, and hindfoot varus and equinus, its causes are multifactorial, involving genetic and environmental factors. Early diagnosis and intervention are essential to prevent lifelong pain and disability. With over 200,000 cases reported annually, the condition often affects both feet but can also present unilaterally, with some populations showing incidence rates as high as 5 per 1,000 births.

The Ponseti method is highly effective for correcting clubfoot initially, though relapse occurs in 30-40% of cases, commonly manifesting as equinus, adductus, or dynamic supination. Factors such as non-compliance with foot abduction orthosis (FAO), incomplete correction, or undiagnosed neuromuscular conditions contribute to relapse. Ensuring parent education, routine follow-ups, and timely bracing adjustments is crucial to reduce these risks.

Treatment options for clubfoot include repeat casting, Achilles tendon lengthening, or tibialis anterior tendon transfer, often avoiding extensive surgery. The Ponseti method, involving weekly manipulations, casting, Achilles tenotomy, Kinesio taping and bracing, achieves up to 98% initial correction but has a 37% relapse rate. Similarly, the French functional method, using manipulations, strapping, and exercises, shows comparable success but also struggles with recurrence.

MFR improves soft tissue flexibility by addressing residual tightness in the foot and lower leg, restoring tissue length, reducing stiffness, and enhancing blood flow for better alignment and functional mobility. Physiotherapy sessions focus on Achilles tendon stretching, mobilization of the tibiotalar, subtalar, and midtarsal joints, and strengthening of the peroneal muscles to promote eversion and stabilization. Proprioceptive exercises, balance training, and functional activities such as weight-bearing and gait training further support motor development. Nighttime bracing maintains the foot in a corrected position, ensuring that soft tissues and joints stay aligned during periods of inactivity.

This integrated approach significantly reduces the risk of relapse, enhances the effectiveness of Ponseti treatment, and improves the child's mobility and quality of life. MFR is a manual therapy technique targeting fascial restrictions to improve mobility, flexibility, and circulation. Fascia, a dense connective tissue surrounding muscles, bones, and organs, can contribute to stiffness and decreased range of motion (ROM) when restricted, increasing the risk of relapse in post-clubfoot treatment Static stretching is commonly used to enhance muscle-tendon flexibility and ROM by modifying passive muscle properties and stretching tolerance. While short-term stretching has limited effects on muscle-tendon unit stiffness (MTS), long-term stretching can significantly reduce stiffness, especially in healthy young individuals. In clubfoot management, static stretching of the gastrocnemius-soleus complex and plantar fascia helps prevent recurrence by maintaining tissue elongation, particularly when combined with nighttime bracing.

The aim of this randomized controlled trial to check the Effect of Myofascial Release and Static Stretching along with Nighttime Bracing in Long-Term Relapse Prevention of Ponseti Treated Clubfoot to optimize long-term mobility, enhance the quality of life for children with idiopathic clubfoot, and reduce the healthcare burden associated with relapse and disability.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with idiopathic clubfoot who have undergone initial correction using Ponseti method.
* The patient is currently in the maintenance (post casting) phase of treatment.
* Age between 0-14 months
* Both unilateral and bilateral
* Children who continue use of bracing for first 3 months
* Both girls and boys

Exclusion Criteria:

* Secondary clubfoot patients
* Cases with a history of non-compliance with Ponseti treatment protocol.
* Children who have the first 3 months on bracing stage

Max Age: 14 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Goniometer | 3 weeks
  To measure ankle range of motion (ROM) with a goniometer, position the patient sitting or lying supine with the knee flexed to 90 degrees. Place the goniometer's axis on the lateral malleolus, aligning the stationary arm with the lateral midline of the fibula and the moving arm parallel to the lateral midline of the fifth metatarsal. For dorsiflexion, pull patient's toes up toward the shin, and record the angle; for plantarflexion, have them point their toes downward, then record the angle.
Pirani Scoring | 3 weeks
  The Pirani score is a standardized clinical tool used to assess the severity of clubfoot deformity, primarily in pediatric patients undergoing Ponseti treatment. It evaluates six specific features across two categories: the midfoot and hindfoot. The midfoot score assesses the medial crease, curvature of the lateral border, and the position of the talus head, with each feature rated from 0 (normal) to 1 (severe), allowing for a maximum of 3 points. The hindfoot score evaluates the posterior crease, rigidity of equines (ankle dorsiflexion limitation), and the "empty heel" sign, with similar scoring criteria. The scores from both categories are combined for a total score ranging from 0 (fully corrected foot) to 6 (most severe deformity).

CONTACTS AND LOCATIONS:
Overall Officials: Hafsa Siddiqui, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Benazir Bhutto Hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No